CLINICAL TRIAL: NCT02554708
Title: pToWin pCONus Treatment of Wide Neck Intracranial Aneurysms
Brief Title: pCONus Treatment of Wide Neck Intracranial Aneurysms
Acronym: pToWin
Status: Completed | Type: Observational
Sponsor: Phenox GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PTW/PV201505-21
Record Dates: First submitted 2015-09-04; First posted 2015-09-18 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Intracranial Aneurysm
Keywords: Aneurysm; bifurcation; wide neck; pCONus; intracerebral; stroke
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: implantation of the pCONus Bifurcation Aneurysm Implant — The device will be introduced through a regular microcatheter. After deployment of the device with the crown positioned in the aneurysm neck the aneurysm will be entered with a microcatheter to perform endovascular coil occlusion. After completion of the coiling procedure the pCONus device will be electrolytically detached from the insertion wire and only the crown and the shaft will remain as a permanent implant.

SUMMARY:
To assess safety and efficacy of pCONus for the treatment of wide neck bifurcation aneurysms.

DETAILED DESCRIPTION:
Title: pCONus Treatment of Wide Neck Intracranial Aneurysms

Acronym: pToWin

Device: pCONus Bifurcation Aneurysm Implant

Study design: Prospective, multicenter, single-arm clinical investigation

Purpose: To assess safety and efficacy of pCONus for the treatment of wide neck bifurcation aneurysms

Duration of the study: 48 months

Sample size: 100 evaluable patients

Number of sites: > 20

Follow-up intervals: Two independent follow-ups (after 3-6 and 7-12 months) according to site specific standard

ELIGIBILITY:
Inclusion Criteria:

1. Aneurysm status:

   * Unruptured aneurysm or
   * Ruptured aneurysm with a Hunt and Hess grade of I - III.
2. Age ≥18 and ≤ 80 years.
3. The patient or legal representative provides written informed consent.
4. The patient shows general compliance to follow the medical regimen and to attend follow-up examinations.
5. The target aneurysm is located at one of the following cerebral vessel bifurcations: ICA terminus, AcomA, MCA or BA.
6. Bifurcation wide neck aneurysm.
7. The dome height should allow for safe deployment of the device crown. The fundus of the aneurysm should offer enough space for the crown of the pCONus to deploy.

Exclusion Criteria:

1. Vessel tortuosity precluding safe access and device deployment.
2. Stenosis within the vascular access or target vessel ≥ 50 %.
3. The target aneurysm has been previously treated with a stent or an intraaneurysmal implant beside coils.
4. The treatment plan for the target aneurysm includes the use of additional intra- and/or extraaneurysmal temporary or permanent implants other than coils.
5. More than one intracerebral aneurysm requires the treatment within the following 6 months.
6. Imaging evidence of an arteriovenous cerebrovascular malformation or a dural fistula.
7. Any physical, medical or psychiatric condition of the patient interfering with the adherence of the requirements and follow-up regimen of the study.
8. Any neurological disorder with progressive neurological symptoms, except attributable to a compressive effect of the target aneurysm.
9. Current involvement in another study or trial.
10. Women of child bearing potential or breast-feeding who cannot provide a negative pregnancy test.
11. Known allergy to the components of device, study medication or contrast media that cannot be controlled medically.
12. A medical condition interfering with a dual antiplatelet treatment.
13. Known coagulopathy.
14. Intracranial hemorrhage in the past 30 days apart from the target aneurysm.
15. Ischemic stroke in the past 30 days.
16. Myocardial infarction in the past 30 days.
17. Major surgery in the past 30 days.
18. Evidence of active infection at time of treatment.
19. Co -morbidities or conditions with a life expectancy less than 12 months.
20. Additional Exclusion criteria for ruptured aneurysm at the acute phase:

    1. The patient is clinically severely affected (Hunt and Hess grade IV and V).
    2. Severe vasospasm is proven during angiography.
    3. Proven parenchymal hemorrhage by CT or MRI.
    4. Proven subdural hematoma by CT or MRI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients harbouring an unruptured or ruptured bifurcation aneurysm, in which pCONus assisted coiling was judged to be the most appropriate treatment
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2015-08; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness Aneurysm occlusion (complete or neck remnant) | Change from post-procedure to 3-6 and to 7-12 months
Safety Major stroke (ischemic or hemorrhagic) or neurological death related to the treatment of the target aneurysm | within 12 months

SECONDARY OUTCOMES:
Effectiveness | at the time of the procedure
  The "Effectiveness endpoint" is assessed throughout the intervention and is assessed as "number/amount of" for each following point:
  * To place pCONus in the desired location
  * Correct opening of the device (crown and shaft)
  * To perform aneurysm occlusion without obliteration of side branches and
  * To detach the device at the end of the procedure
Safety Intra-Procedural Complications | at the time of the procedure
  The "Safety Intra-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of" for each following point:
  * Vessel perforation
  * Target aneurysm perforation with microcatheter or guidewire
  * Target aneurysm perforation with pCONus
  * Target aneurysm perforation with coils
  * Thromboembolism
  * Dissection of any access vessel
Safety Post-Procedural Complications | Change 1day post procedure up to 12months
  The "Safety Post-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of" for each following point:
  * Frequency of new parenchymal hemorrhage during the follow-up period
  * Frequency of new subarachnoid hemorrhage during the follow-up period
  * Frequency of new ischemic stroke on follow-up imaging
  * Rupture of the target aneurysm during the 12 months follow-up period
  * Rate of in-stent-stenosis
  * Rate of in-stent-thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Biondi, Prof. Dr., Principal Investigator — Hôpital Jean Minjoz (CHU Besançon), France
Locations (10):
- Clínica La Sagrada Familia Department of Neuroscience (P.L.), Equipo de Neurocirugía Endovascular y Radiología Intervencionista, Buenos Aires, Buenos Aires F.D., Argentina
- LKH-Univ. Klinikum Graz Universitätsklinik für Radiologie, Graz, Austria
- Hôpital Pierre Wertheimer (HCL Groupement Hospitalier Est), Bron, France
- Germany (6):
  - KRH Klinikum Nordstadt, Hanover, Lower Saxony
  - Universitätsklinikum Heidelberg, Heidelberg
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Koblenz
  - Klinikum Osnabrück, Osnabrück
  - Knappschaftskrankenhaus Recklinghausen, Recklinghausen
  - Klinikum Stuttgart Katharinenhospital, Stuttgart
- A.S.L. Napoli 1 Centro - P.O. San Giovanni Bosco, Napoli, Italy

REFERENCES:
- [Background] Aguilar Perez M, Henkes H, Kurre W, Bleise C, Lylyk PN, Lundquist J, Turjman F, Alhazmi H, Loehr C, Felber S, Deutschmann H, Lowens S, Delehaye L, Mohlenbruch M, Hattingen J, Lylyk P. Results of the pToWin Study: Using the pCONUS Device for the Treatment of Wide-Neck Intracranial Aneurysms. J Clin Med. 2022 Feb 8;11(3):884. doi: 10.3390/jcm11030884. PMID 35160333